CLINICAL TRIAL: NCT00159913
Title: A Randomized, Double-Blind, Placebo Controlled, Dose Ranging, Parallel Group Study of Oral Sildenafil in the Treatment of Children, Aged 1-17 Years, With Pulmonary Arterial Hypertension.
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study of Sildenafil in Children With Pulmonary Arterial Hypertension.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A1481131
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Arterial Hypertension, Children
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sildenafil Low dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil Medium dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Sildenafil High dose (Experimental)
  Interventions: Drug: Sildenafil citrate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil citrate — oral; 20mg, 40mg and 80 mg; 3 times a day(TID)
  Arms: Sildenafil High dose
Drug: Sildenafil citrate — oral; 10mg, 20mg and 40mg; 3 times a day(TID)
  Arms: Sildenafil Medium dose
Drug: Placebo — oral; 3 times a day(TID)
  Arms: Placebo
Drug: Sildenafil citrate — oral; 10 mg; 3 times a day(TID)
  Arms: Sildenafil Low dose

SUMMARY:
This is a clinical research study designed to evaluate sildenafil for the treatment of Pulmonary Arterial Hypertension in children, aged 1 to 17 years. The purpose of the study is to assess the efficacy, safety, and pharmacokinetics of 16 weeks of chronic treatment with oral sildenafil given in three different doses, compared to placebo (inactive treatment). Efficacy will be measured by exercise and hemodynamics. Patients who complete this trial may be eligible to take part in an extension study, in which all patients will receive active treatment of sildenafil.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged from 1 to 17 years old and weighing >= 8 kg with a mean pulmonary artery pressure >= 25 mmHg at rest, PCWP <= 15 mmHg, and PVRI >= 3 Wood units x m2 (if PCWP is not available, then mean LA pressure <= 15 mmHg or LVEDP <= 15 mmHg in the absence of left atrial obstruction).
* Females of child bearing potential who were sexually active must have been practicing a suitable method of birth control so that in the opinion of the investigator, they would not become pregnant during the study.
* Subjects who have symptomatic pulmonary arterial hypertension due to: primary pulmonary hypertension; pulmonary arterial hypertension in the presence of a small or hemodynamically insignificant congenital systemic to pulmonary shunt lesion that in the opinion of the investigator is not the cause of pulmonary hypertension; collagen vascular disease; congenital systemic-to-pulmonary shunts with a baseline resting room air oxygen saturation >= 88% unrepaired or repaired at least 6 months prior to screening; d-transposition of the great arteries repaired within the first 30 days of life; or surgical repair of other congenital heart lesions at least 6 months prior to screening and do not have clinically significant residual left-sided heart disease consistent with the exclusion criteria.
* Subjects, developmentally able to exercise, whose CPX exercise test functional capacity is within the following parameters: Peak VO2 >= 10 mL/kg/min and <= 28 mL/kg/min during screening CPX test;
* Written informed consent and assent where applicable before the subject is screened for the study.
* Subjects who undergo a large shift in altitude (defined as approximately 5000 feet or 1524 meters) in order to participate in the study must reside at the "in study" altitude for at least 90 days prior to baseline and during the study period.

Exclusion Criteria:

* Subjects with pulmonary hypertension secondary to sickle cell disease, any other disease known to be associated with PAH, or any etiology other than those specified in the inclusion criteria.
* Left-sided heart disease, including aortic or mitral valve disease (greater than mild), restrictive or congestive cardiomyopathy; PCWP or LVEDP > 15 mmHg; LVEF < 40% determined by MUGA, angiography or echocardiography; LV shortening fraction < 22% determined by echocardiography, symptomatic coronary disease (demonstrable ischemia).
* Pericardial constriction; significant (2+ for regurgitation) valvular disease other than tricuspid or pulmonary regurgitation; acutely decompensated heart failure within previous 30 days from screening; atrial septostomy within previous 6 months of screening;
* Hemodynamic instability or hypo- or hypertension at screening, i.e., SBP outside of 70-140 mmHg.
* A history of stroke, myocardial infarction or life threatening arrhythmia within 6 months of screening.
* Moderate to severe restrictive pulmonary disease (Total Lung Capacity or Forced Vital Capacity <= 60% of normal) or history of severe lung disease.
* Subjects with bronchopulmonary dysplasia (BPD) and other chronic lung diseases.
* History of pulmonary embolism.
* Subjects whose CPX test is limited by conditions other than pulmonary hypertension-associated dyspnea or fatigue.
* Subjects who are known to be HIV positive
* Subjects with impairment of renal function (serum creatinine > 2.5x ULN ) or hepatic function (ALT and/or AST > 3x ULN; and/or bilirubin >= 2 mg/dL). Hematological abnormalities (e.g., severe anemia, Hgb < 10 g/dL, leukopenia, WBC < 2500/mL).
* Subjects who previously received bosentan and whose liver function tests taken at screening are > 2x ULN.
* Subjects with any medical condition which in the opinion of the investigator may interfere with treatment, evaluation of safety, and/or efficacy.
* Change in class of medication for CHF or PAH within the 10 days prior to qualifying right heart catheterization.
* Subjects who are currently prescribed and/or taking nitrates or nitric oxide donors in any form. Acute vasodilator testing with nitric oxide is permitted during hemodynamic evaluation; taking chronic arginine supplementation including Heart Bar; therapy involving parenteral inotropic medication or parenteral vasodilators within 3 months of screening; current therapy with alpha-blockers, potent cytochrome P450 3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole and protease inhibitors), Ritonavir or Nicorandil; chronic treatment with off-label sildenafil, an endothelin antagonist or prostacyclin/prostacyclin analogue within 30 days of randomization.
* Pregnant or lactating female.
* Any medical or psychological condition or social circumstances that would impair their ability to participate reliably in the study or who were not likely to complete the study for any reason; current or past illicit drug use or alcoholism excepting if abstinence can be documented for >= 1 year.
* Participation in another clinical trial of an investigational drug or device (including placebo) within 30 days of screening for entry into the present study.
* Subjects with known hereditary degenerative retinal disorders (such as retinitis pigmentosa) or history of non-arteritic anterior ischemic optic neuropathy (NAION).

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 235 (Actual)
Dates: Start 2003-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (34):
- United States (10):
  - Pfizer Investigational Site, Palo Alto, California
  - Pfizer Investigational Site, Stanford, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Seattle, Washington
- Pfizer Investigational Site, São Paulo, São Paulo, Brazil
- Pfizer Investigational Site, Edmonton, Alberta, Canada
- Pfizer Investigational Site, Santiago, RM, Chile
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogota, Cundinamarca
- Pfizer Investigational Site, Guatemala City, Guatemala
- Hungary (3):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Deszk
  - Pfizer Investigational Site, Szeged
- India (2):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Kerala, Kochi,
- Pfizer Investigational Site, Bologna, Italy
- Pfizer Investigational Site, Tokyo, Japan
- Pfizer Investigational Site, George Town, Pulau Pinang, Malaysia
- Mexico (2):
  - Pfizer Investigational Site, Del. Tlalpan, Mexico City
  - Pfizer Investigational Site, Tlalpan, Mexico DF
- Pfizer Investigational Site, Lima, Peru
- Poland (3):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze
- Pfizer Investigational Site, Moscow, Russia
- Pfizer Investigational Site, Lund, Sweden
- Taiwan (2):
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei

REFERENCES:
- [Derived] Russell S, Beghetti M, Oudiz R, Balagtas C, Zhang M, Ivy D. Effects of oral sildenafil on exercise capacity in children with pulmonary arterial hypertension: a randomised trial. Open Heart. 2019 Dec 3;6(2):e001149. doi: 10.1136/openhrt-2019-001149. eCollection 2019. PMID 31908813
- [Derived] Chanu P, Gao X, Bruno R, Claret L, Harnisch L. A modeling and simulation-based assessment of the impact of confounding factors on the readout of a sildenafil survival trial in pulmonary arterial hypertension. J Pharmacokinet Pharmacodyn. 2019 Oct;46(5):499-509. doi: 10.1007/s10928-019-09654-3. Epub 2019 Sep 20. PMID 31538282
- [Derived] Beghetti M, Rudzinski A, Zhang M. Efficacy and safety of oral sildenafil in children with Down syndrome and pulmonary hypertension. BMC Cardiovasc Disord. 2017 Jul 4;17(1):177. doi: 10.1186/s12872-017-0569-3. PMID 28676038
- [Derived] Cappelleri JC, Hwang LJ, Mardekian J, Mychaskiw MA. Assessment of measurement properties of peak VO(2) in children with pulmonary arterial hypertension. BMC Pulm Med. 2012 Sep 10;12:54. doi: 10.1186/1471-2466-12-54. PMID 22963001
- [Derived] Barst RJ, Ivy DD, Gaitan G, Szatmari A, Rudzinski A, Garcia AE, Sastry BK, Pulido T, Layton GR, Serdarevic-Pehar M, Wessel DL. A randomized, double-blind, placebo-controlled, dose-ranging study of oral sildenafil citrate in treatment-naive children with pulmonary arterial hypertension. Circulation. 2012 Jan 17;125(2):324-34. doi: 10.1161/CIRCULATIONAHA.110.016667. Epub 2011 Nov 29. PMID 22128226
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481131&StudyName=A%20Randomized%2C%20Double-Blind%2C%20Placebo-Controlled%20Study%20of%20Sildenafil%20in%20Children%20with%20Pulmonary%20Arterial%20Hypertension.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 centers in North, Latin and South America, Europe and Asia.
Pre-assignment Details: Of the 324 subjects screened, 235 subjects were randomized. 234 received treatment. One subject(sildenafil medium dose group) withdrew prior to taking any study treatment as the hemodynamic entrance criteria were not met.
Groups:
- Sildenafil Low Dose: Day 1-7 10 mg, followed by 10 mg TID (3 times daily) for body weights > 20-45 kg and > 45 kg, through Day 112.
  Modeling of the plasma concentrations for each dose level showed that the low and medium doses were predicted to be similar for the 8 to 20 kg subjects (ie, subjects would receive the same dose because of the available tablet strengths); consequently there was no low dose for the >= 8-20 kg weight group.
- Sildenafil Medium Dose: Day 1-7 10 mg, followed by 10, 20, 40 mg TID (3 times daily) for body weights >= 8-20 kg, > 20-45 kg, > 45 kg respectively, through Day 112
- Sildenafil High Dose: Day 1-7 10 mg, followed by 20, 40, 80 mg TID (3 times daily) for body weights >= 8-20 kg, > 20-45 kg, > 45 kg respectively, through Day 112
- Placebo: Subjects randomized to this arm recieved placebo TID (three times daily) for 112 days.
Period: Overall Study
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Placebo
Started | 42 | 55 | 77 | 60
Completed | 40 | 55 | 75 | 58
Not Completed | 2 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Placebo | Total
Number analyzed (Participants) | 42 | 55 | 77 | 60 | 234
Age, Customized [Number; unit: participants]
  1-4 Years | 0 | 9 | 19 | 7 | 35
  5-12 Years | 25 | 28 | 36 | 37 | 126
  13-17 Years | 17 | 18 | 22 | 16 | 73
  >= 18 Years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 31 | 51 | 38 | 145
  Male | 17 | 24 | 26 | 22 | 89

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Peak Volume of Oxygen (VO2) Consumed : Intent To Treat Population
Description: Peak VO2 (normalized for body weight) at trough plasma levels assessed by CPX testing (bicycle ergometry)at the end of treatment (Week 16 for those who completed the study). Mean Percent change = [(week 16 value minus baseline mean)/mean at baseline]*100%.
Time Frame: Baseline, Week 16
Population: ITT population included all subjects randomised and who received at least one dose of study medication. All subjects developmentally able to perform the exercise test. Subjects assumed developmentally able if they had a CPX exercise assessment at any visit during study using a LOCF (end-of-treatment)approach for handling missing data.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Combined Sildenafil: This includes all subjects in the low, medium and high dose groups.
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 24 | 26 | 27 | 77 | 29
percent change | 6.44 (20.16) [-6.11 to 13.73] | 13.40 (19.50) [1.72 to 20.94] | 10.58 (15.51) [-1.64 to 17.60] | 10.24 (18.39) | 0.53 (15.91)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA — No adjustments for multiple comparisons have been made; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Net) = 7.71, 95% CI [-0.19 to 15.60], Standard Error of Mean 3.98
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Net) = 3.81, 95% CI [-6.11 to 13.73], Standard Error of Mean 5.00
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Net) = 11.33, 95% CI [1.72 to 20.94], Standard Error of Mean 4.84
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Net) = 7.98, 95% CI [-1.64 to 17.60], Standard Error of Mean 4.85

2. Secondary Outcome: Change From Baseline to Week 16 in Mean Pulmonary Artery Pressure (mPAP)
Description: mPAP, a hemodynamic parameter, was measured using a pressure transducer positioned at the mid-axillary line with the patient in the supine position. Change is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, using a LOCF (end-of-treatment) approach for handling missing data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 39 | 55 | 71 | 165 | 56
mm Hg | 0.9 (12.3) | -3.9 (12.0) | -7.4 (15.4) | -4.3 (13.9) | -0.4 (15.9)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.172, ANCOVA; Covariates:etiology, wt grp, capability performing exercise test. Normality assumptions not met with main analysis: alternative=excluding outliers; Mean Difference (Final Values) = -3.1, 95% CI [-7.5 to 1.3], Standard Error of Mean 2.2
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 1.6, 95% CI [-4.5 to 7.6], Standard Error of Mean 3.1
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI [-8.9 to 1.9], Standard Error of Mean 2.7
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -7.3, 95% CI [-12.4 to -2.1], Standard Error of Mean 2.6

3. Secondary Outcome: Change From Baseline to Week 16 in Pulmonary Vascular Resistance Index (PVRI)
Description: PVRI equals Pulmonary Vascular Resistance (PVR) times Body Surface Area (BSA). Wood unit = 80dyn•s/cm5. Change is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, LOCF
Measure: Mean (Standard Deviation); unit: wood units. m2
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 36 | 49 | 67 | 152 | 50
wood units. m2 | 0.1 (10.9) | -2.9 (11.5) | -5.1 (14.7) | -3.2 (13.0) | 1.6 (9.2)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.041, ANCOVA; Covariates:etiology, wt grp, capability performing exercise test. Normality assumptions not met w/ main analysis: alternative=natural log transformed; Mean Difference (Final Values) = -4.1, 95% CI [-8.0 to -0.2], Standard Error of Mean 2.0
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI [-5.9 to 4.7], Standard Error of Mean 2.7
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.5, 95% CI [-9.3 to 0.3], Standard Error of Mean 2.4
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.2, 95% CI [-11.7 to -2.7], Standard Error of Mean 2.3

4. Secondary Outcome: Percent Change From Baseline to Week 16 in: Respiratory Exchange Ratio (RER)
Description: RER is the ratio of carbon dioxide produced to oxygen consumed [VCO2/VO2]). Percent change is [(Week 16 value minus Baseline value)/Baseline value] * 100%
Time Frame: Baseline, Week 16
Population: ITT population, LOCF (end-of-treatment) approach for handling missing values.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 24 | 26 | 27 | 77 | 29
percent change | -0.00 (0.13) | -0.05 (0.12) | -0.02 (0.11) | -0.03 (0.12) | -0.03 (0.11)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.795, ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 0.61, 95% CI [-4.07 to 5.30], Standard Error of Mean 2.36
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 2.62, 95% CI [-3.31 to 8.54], Standard Error of Mean 2.99
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = -1.29, 95% CI [-7.09 to 4.50], Standard Error of Mean 2.92
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 0.52, 95% CI [-5.24 to 6.28], Standard Error of Mean 2.90

5. Secondary Outcome: Percent Change From Baseline to Week 16 in Time to Maximum Volume of Oxygen Consumed (VO2)
Description: Time to maximum VO2 was assessed on the subset of subjects who are developmentally able to perform the exercise test. Percent change is [(value at Week 16 minus Baseline value)/Baseline value] * 100%
Time Frame: Baseline, Week 16
Population: ITT population, LOCF (end-of-treatment) approach for handling missing values.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 24 | 26 | 27 | 77 | 29
percent change | 64.83 (103.69) | 64.42 (102.70) | 31.33 (107.04) | 52.95 (104.40) | 8.84 (96.09)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.139, ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 9.24, 95% CI [-3.05 to 21.54], Standard Error of Mean 6.20
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 10.34, 95% CI [-5.21 to 25.90], Standard Error of Mean 7.84
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 11.43, 95% CI [-3.78 to 26.64], Standard Error of Mean 7.67
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology and weight group; Mean Difference (Final Values) = 5.96, 95% CI [-9.16 to 21.08], Standard Error of Mean 7.62

6. Secondary Outcome: Change From Baseline to Week 16 in Pulmonary Vascular Resistance (PVR)
Description: Change calculated as (mean PAP - PCWP)/COpulm in PVR is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, using LOCF (end of treatment) approach for handling missing data
Measure: Mean (Standard Deviation); unit: wood units
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 36 | 49 | 67 | 152 | 50
wood units | -0.1 (10.4) | -3.3 (10.5) | -5.2 (15.7) | -3.4 (13.1) | 0.1 (11.8)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.172, ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -2.9, 95% CI [-7.1 to 1.3], Standard Error of Mean 2.1
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = 0.2, 95% CI [-5.5 to 5.9], Standard Error of Mean 2.9
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -3.4, 95% CI [-8.5 to 1.7], Standard Error of Mean 2.6
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -5.5, 95% CI [-10.3 to -0.7], Standard Error of Mean 2.4

7. Secondary Outcome: Change From Baseline to Week 16 in Cardiac Index (CI)
Description: CI is observed value at Week 16 minus Baseline value. Calculated as cardiac output in systemic circulation (COsys) / body surface area (BSA).
Time Frame: Baseline, Week 16
Population: ITT population, using LOCF (end of treatment) approach for handling missing data.
Measure: Mean (Standard Deviation); unit: liters/minute/meters squared
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 37 | 49 | 68 | 154 | 52
liters/minute/meters squared | 0.20 (1.17) | 0.02 (1.44) | 0.24 (2.19) | 0.16 (1.76) | -0.60 (2.12)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = 0.74, 95% CI [0.14 to 1.34], Standard Error of Mean 0.30
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = 0.71, 95% CI [-0.10 to 1.52], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = 0.61, 95% CI [-0.12 to 1.35], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = 0.89, 95% CI [0.21 to 1.58], Standard Error of Mean 0.35

8. Secondary Outcome: Change From Baseline to Week 16 in Right Atrial Pressure (RAP)
Description: RAP was measured using a pressure transducer positioned at the mid-axillary line with the patient in the supine position. Change is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, using LOCF (end of treatment) approach for missing data.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 39 | 55 | 71 | 165 | 56
mm Hg | 7.92 (2.85) | 8.05 (4.42) | 7.75 (4.14) | 7.89 (3.95) | 8.11 (3.61)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.440, ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -0.50, 95% CI [-1.77 to 0.77], Standard Error of Mean 0.64
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -0.17, 95% CI [-1.91 to 1.57], Standard Error of Mean 0.88
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -0.19, 95% CI [-1.73 to 1.36], Standard Error of Mean 0.78
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; The model included the covariates etiology, weight group and capability of performing the exercise test; Mean Difference (Final Values) = -1.14, 95% CI [-2.61 to 0.33], Standard Error of Mean 0.75

9. Secondary Outcome: Change From Baseline to Week 16 in Child Health Questionnaire Parent Form (CHQ-PF28), Physical Scale
Description: CHQ-PF28: validated generic Quality of Life (QoL) questionnaire for subjects >= 5 years. Includes 12 domain scores of QoL concepts including physical functioning, social & school activities, mental health, parent/family concepts. Scores range 0-100: lower scores = lower QoL. Change is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, includes subjects >= 5 years with a valid questionnaire available in the subject's first language.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 31 | 29 | 43 | 103 | 40
score on scale | 14.0 (13.1) | 9.8 (11.8) | 5.9 (10.5) | 9.4 (12.1) | 8.3 (12.0)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.750, ANCOVA; The covariates included in the model were baseline scale, etiology, weight and capability of performing the exercise test; Mean Difference (Final Values) = -0.62, 95% CI [-4.45 to 3.21], Standard Error of Mean 1.93
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.87, 95% CI [-4.21 to 5.95], Standard Error of Mean 2.57
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.24, 95% CI [-4.68 to 5.15], Standard Error of Mean 2.49
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -2.96, 95% CI [-7.37 to 1.45], Standard Error of Mean 2.23

10. Secondary Outcome: Change From Baseline to Week 16 in Child Health Questionnaire Parent Form (CHQ-PF28), Psychosocial Scales
Description: as for outcome 9
Time Frame: Baseline, Week 16
Population: ITT population, includes subjects >= 5years with a valid questionnaire available in the subject's first language.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 34 | 30 | 45 | 109 | 41
score on scale | 5.1 (6.9) | 4.1 (8.1) | 4.3 (10.0) | 4.5 (8.6) | 5.6 (10.3)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.784, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI [-3.41 to 2.58], Standard Error of Mean 1.51
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.41, 95% CI [-3.49 to 4.30], Standard Error of Mean 1.97
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -2.11, 95% CI [-5.99 to 1.77], Standard Error of Mean 1.96
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.46, 95% CI [-3.06 to 3.97], Standard Error of Mean 1.77

11. Secondary Outcome: Change From Baseline to Week 16 in World Health Organization (WHO) Pulmonary Hypertension (PH) Functional Class
Description: WHO PH functional class definitions adapted from New York Heart Association Criteria for Functional Capacity and Therapeutic Class Definitions. Class I = PH without resulting limitation of physical activity, Class II = PH resulting in slight limitation of physical activity, Class III = PH resulting in marked limitation of physical activity, Class IV = PH with inability to carry out any physical activity without symptoms. Improved by 1 class = Class 4 to 3, Class 3 to 2, Class 2 to 1. Improved by 2 classes = Class 4 to 2, Class 3 to 1. Change is observed value at Week 16 minus Baseline value.
Time Frame: Baseline, Week 16
Population: ITT population, LOCF
Measure: Number; unit: units
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 31 | 34 | 55 | 120 | 35
units
  No change | 25 | 24 | 38 | 84 | 31
  Improved by 1 class | 6 | 10 | 16 | 32 | 4
  Improved by 2 classes | 0 | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.184, Regression, Logistic; Proportional odds method. Model covariates were baseline WHO functional class, etiology, weight group and capability of performing the exercise test; Odds Ratio (OR) = 1.83, 95% CI [0.75 to 4.45]
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; p = 0.409, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 0.60, 95% CI [0.18 to 2.01]
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; p = 0.146, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 2.25, 95% CI [0.75 to 6.69]
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; p = 0.006, Regression, Logistic; [statistical method as in outcome 11, analysis 1]; Odds Ratio (OR) = 4.52, 95% CI [1.56 to 13.10]

12. Primary Outcome: Percent Change From Baseline in Peak Volume of Oxygen (VO2) Consumed : Per Protocol Population
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Number analyzed (Participants) | 23 | 23 | 27 | 73 | 24
percent change | 5.43 (20.69) | 15.66 (21.48) | 9.34 (17.13) | 10.10 (19.87) | 2.81 (13.17)
Statistical Analysis 1: Comparison: Combined Sildenafil vs Placebo; Test type: Superiority or Other; p = 0.179, ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Final Values) = 5.89, 95% CI [-2.74 to 14.53], Standard Error of Mean 4.35
Statistical Analysis 2: Comparison: Sildenafil Low Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Final Values) = 1.14, 95% CI [-9.49 to 11.77], Standard Error of Mean 5.35
Statistical Analysis 3: Comparison: Sildenafil Medium Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Final Values) = 11.30, 95% CI [0.66 to 21.96], Standard Error of Mean 5.36
Statistical Analysis 4: Comparison: Sildenafil High Dose vs Placebo; Test type: Superiority or Other; ANCOVA; Analyses performed using analysis of covariance with etiology, weight and baseline peak VO2 as the covariates; Mean Difference (Final Values) = 5.24, 95% CI [-5.02 to 15.50], Standard Error of Mean 5.16

ADVERSE EVENTS:
Arm/Group | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 7 | 9 | 2
Other Adverse Events (participants affected / at risk) | 22 | 37 | 44 | 102 | 29
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Bradycardia (Cardiac disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Cardiac failure congestive (Cardiac disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Cyanosis (Cardiac disorders) | 1/42 | 0/55 | 0/77 | 1/174 | 0/60
Ventricular arrhythmia (Cardiac disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Diarrhoea (Gastrointestinal disorders) | 0/42 | 0/55 | 0/77 | 0/174 | 1/60
Haematochezia (Gastrointestinal disorders) | 1/42 | 0/55 | 0/77 | 1/174 | 0/60
Pyrexia (General disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Gastroenteritis (Infections and infestations) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Pneumonia (Infections and infestations) | 0/42 | 1/55 | 2/77 | 3/174 | 0/60
Pneumonia bacterial (Infections and infestations) | 0/42 | 0/55 | 0/77 | 0/174 | 1/60
Upper respiratory tract infection (Infections and infestations) | 0/42 | 1/55 | 1/77 | 2/174 | 0/60
Syncope (Nervous system disorders) | 1/42 | 0/55 | 0/77 | 1/174 | 0/60
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/42 | 0/55 | 0/77 | 1/174 | 0/60
Stridor (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/55 | 1/77 | 1/174 | 0/60
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sildenafil Low Dose | Sildenafil Medium Dose | Sildenafil High Dose | Combined Sildenafil | Placebo
Anaemia (Blood and lymphatic system disorders) | 0/42 | 2/55 | 0/77 | 2/174 | 1/60
Conjunctivitis (Eye disorders) | 0/42 | 0/55 | 2/77 | 2/174 | 2/60
Abdominal pain (Gastrointestinal disorders) | 1/42 | 0/55 | 2/77 | 3/174 | 3/60
Abdominal pain lower (Gastrointestinal disorders) | 0/42 | 0/55 | 3/77 | 3/174 | 0/60
Abdominal pain upper (Gastrointestinal disorders) | 0/42 | 3/55 | 3/77 | 6/174 | 1/60
Diarrhoea (Gastrointestinal disorders) | 2/42 | 3/55 | 7/77 | 12/174 | 4/60
Dyspepsia (Gastrointestinal disorders) | 0/42 | 2/55 | 0/77 | 2/174 | 1/60
Nausea (Gastrointestinal disorders) | 0/42 | 4/55 | 4/77 | 8/174 | 0/60
Vomiting (Gastrointestinal disorders) | 3/42 | 5/55 | 11/77 | 19/174 | 4/60
Chest pain (General disorders) | 2/42 | 1/55 | 2/77 | 5/174 | 2/60
Fatigue (General disorders) | 2/42 | 0/55 | 2/77 | 4/174 | 1/60
Bronchitis (Infections and infestations) | 2/42 | 5/55 | 3/77 | 8/174 | 1/60
Influenza (Infections and infestations) | 0/42 | 2/55 | 0/77 | 2/174 | 0/60
Laryngitis (Infections and infestations) | 1/42 | 0/55 | 1/77 | 2/174 | 2/60
Nasopharyngitis (Infections and infestations) | 3/42 | 3/55 | 2/77 | 8/174 | 4/60
Pharyngitis (Infections and infestations) | 3/42 | 3/55 | 1/77 | 7/174 | 0/60
Pneumonia (Infections and infestations) | 0/42 | 2/55 | 0/77 | 2/174 | 0/60
Rhinitis (Infections and infestations) | 1/42 | 3/55 | 1/77 | 5/174 | 1/60
Upper respiratory tract infection (Infections and infestations) | 4/42 | 8/55 | 6/77 | 18/174 | 4/60
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2/42 | 0/55 | 0/77 | 2/174 | 2/60
Dizziness (Nervous system disorders) | 2/42 | 2/55 | 2/77 | 6/174 | 2/60
Headache (Nervous system disorders) | 5/42 | 6/55 | 12/77 | 23/174 | 8/60
Enuresis (Renal and urinary disorders) | 0/42 | 2/55 | 0/77 | 2/174 | 0/60
Erection increased (Reproductive system and breast disorders) | 0/42 | 1/55 | 2/77 | 3/174 | 0/60
Spontaneous penile erection (Reproductive system and breast disorders) | 0/42 | 2/55 | 1/77 | 3/174 | 0/60
Cough (Respiratory, thoracic and mediastinal disorders) | 2/42 | 4/55 | 2/77 | 8/174 | 3/60
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/42 | 2/55 | 3/77 | 6/174 | 2/60
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/42 | 2/55 | 0/77 | 3/174 | 1/60
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/42 | 0/55 | 0/77 | 0/174 | 2/60
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/42 | 4/55 | 2/77 | 6/174 | 0/60
Rash macular (Skin and subcutaneous tissue disorders) | 0/42 | 2/55 | 1/77 | 3/174 | 0/60
Flushing (Vascular disorders) | 1/42 | 1/55 | 0/77 | 2/174 | 3/60
Pyrexia (General disorders) | 3/42 | 8/55 | 8/77 | 19/174 | 1/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.